CLINICAL TRIAL: NCT00805272
Title: Medical and Economical Evaluation of New Diagnosis Tests of Mycobacterium Tuberculosis, Specific Immune Responses in HIV-infected Adults
Brief Title: Medical and Economical Impact of IGRAs Diagnosis of Latent Tuberculosis in HIV-infected Patients
Acronym: IGRAVIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P070311
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2008-11

CONDITIONS: HIV; Tuberculosis; Latent Tuberculosis Infection
Keywords: HIV; tuberculosis; IGRA; diagnosis; treatment naive
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Other: QTF-TB Gold and T-SPOT TB

INTERVENTIONS:
Other: QTF-TB Gold and T-SPOT TB — evaluation of the theoric therapeutic impact of the use of IGRAS for diagnosis of LTBI in HIV-infected patients
  Other Names: IGRAVIH

SUMMARY:
Tuberculosis is a current infection during HIV infection. After infectious contact, some patients will develop tuberculosis some will only be infected without symptoms, they have Latent Tuberculosis Infection (LTBI) which can reactivate later.In order to prevent this tuberculosis reactivation, LTBI diagnosis screening is preconised in HIV-infected patients. This diagnosis is made till now by the tuberculin skin test (TST) but this test is not specific of TB. New blood tests (QFTB-G and T-SPOT.TB) specific po MTB infection are now sold but have not been evaluated in immunocompromised HIV-infected patients.

The primary endpoint of this study is the evaluation of the theoretic therapeutic impact of the use of IGRAS for diagnosis of LTBI in HIV-infected patients

DETAILED DESCRIPTION:
Principal outcome:

-Theoretic therapeutic impact evaluation of the use of IGRAS for diagnosis of LTBI in HIV-infected patients .

Secondary outcomes:

* Medico-economic impact of replacement of TST by IGRAs in LTBI screening in HIV infected patients.
* Concordance of IGRAs results with TST
* Concordance between IGRAs.
* Concordance between IGRAs in accordance to CD4 number(< 100, 100 à 200, 200 à 300, > à 300/mm3).
* LTBI prevalence in the study group.
* Effective consequences of tests results on therapeutic outcome of the patients LTBI criteria and therapeutic recommendations
* One or 2 positive IGRAs test: LTBI recommended to be LTBI
* 1 negative IGRAs test and one undetermined : no LTBI
* 2 undetermined:
* No clinical risk and negative TST: no diagnosis, eventually new test at 3 months or after HAART onset.
* Clinical risk or TST> 10mm: LTBI recommended to be treated. Therapeutic outcome evaluation Effective consequences of IGRA's result on patients outcome at 6 months.

Analyzed criteria:

Therapeutic impact:

* Patients percentage with different therapeutic outcome based on usual recommendations
* Medico-economic impact
* Medico-economic impact of both tests as early and late cost - efficacy
* Statistics

Primary criteria:

* Percentage of patients for whom therapeutic would have been changed by IGRAs results compared to usual diagnosis strategy.

Secondary criteria:

* Concordance of IGRAs with TST
* Concordance between both IGRAs.
* Taille: 1000 patients

Timing:

-inclusions: 2 years

ELIGIBILITY:
Inclusion Criteria:

18 yrs old Confirmed HIV infection No HAART Consent signed 6 months follow-up possible

Exclusion Criteria:

Confirmed TB disease No social right pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2009-02; Primary Completion 2011-09 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the theoretical therapeutic impact (in terms of CHIMIOPROPHYLAXIE antituberculous theoretically managed) of the tracking of tuberculosis-latent by QTF-TB Gold IT® or T-SPOT.TB among patients HIV. | J0

CONTACTS AND LOCATIONS:
Overall Officials: BOURGARIT Anne, Principal Investigator — APHP
Locations (1):
- Service de médecine interne hôpital saint louis, Paris, Paris, France

REFERENCES:
- [Derived] Bourgarit A, Baron G, Breton G, Tattevin P, Katlama C, Allavena C, Campa P, Ravaud P, Lortholary O, Carcelain G; IGRAVIH Study Group. Latent Tuberculosis Infection Screening and 2-Year Outcome in Antiretroviral-Naive HIV-Infected Patients in a Low-Prevalence Country. Ann Am Thorac Soc. 2015 Aug;12(8):1138-45. doi: 10.1513/AnnalsATS.201412-600OC. PMID 26213798